CLINICAL TRIAL: NCT02518477
Title: LYCA: Preventive Intervention Against Lymphedema After Breast Cancer Surgery - a Randomized Controlled Trial
Brief Title: Preventive Intervention Against Lymphedema After Breast Cancer Surgery
Acronym: LYCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Cancer Society (Other)
Collaborators: Rigshospitalet, Denmark (Other); Herlev Hospital (Other); Ringsted sygehus (Unknown)
Responsible Party: Principal Investigator, Oksbjerg Dalton, MD PhD, Danish Cancer Society
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R96-A6604-14-S22
Record Dates: First submitted 2015-08-04; First posted 2015-08-07 (Estimated); Last update posted 2018-09-14 (Actual); Status verified 2018-09

CONDITIONS: Breast Neoplasms
Keywords: breast cancer surgery; axillary lymph node dissection; resistance training; breast cancer related lymphedema
MeSH Terms: conditions — Breast Neoplasms; Breast Cancer Lymphedema | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- exercise group (Experimental): The first 20 weeks, twice-weekly 60 minute session of physical exercise supervised by the research assistant and once weekly home exercise programme is offered. The exercise intervention will consist of stretching, scar tissue mobilization and resistance exercises.
  For the following 32 weeks a home-training manual specifying three times weekly training is provided. At week 26 an individual booster session will be offered. In the case of lymphedema, referral to trained lymphedema physiotherapist for evaluation of appropriate intervention is made.
  Interventions: Other: exercise
- usual care control group (No Intervention): Receives all standard care offered from the operating hospital and rehabilitation in the municipality.

INTERVENTIONS:
Other: exercise — progressive resistance training
  Arms: exercise group

SUMMARY:
This study will examine whether lymphedema after breast cancer surgery can be reduced. In a randomised controlled design the aim is to investigate whether an early intervention with progressive resistance training and close monitoring of arm swelling can reduce the incidence of lymphedema after breast cancer surgery.

DETAILED DESCRIPTION:
Lymphedema is a well known and much dreaded complication after breast cancer surgery. The aim in this study is to examine if lymphedema can be prevented with early progressive strength training focusing on the arm, and close monitoring of pre clinical lymphedema in the 1 year exercise period. The primary outcome is lymphedema, and secondary outcomes are pain, self-reported symptoms of swelling, sensory disturbance, physical and psychological functioning, fatigue, depression, anxiety and health related quality of life.

158 patients operated for breast cancer with axillary node dissection, will be invited from three hospitals in Denmark, Sealand (Rigshospitalet, Ringsted Hospital, and Herlev Hospital), while on the surgical wards. Two weeks later upon consent they are recruited, baseline tested and randomized to either exercise intervention or usual care control.

The exercise intervention consists of progressive resistance training, combined with a stretching programme, with a total duration of 60 minutes per session. The group attend supervised exercises twice a week and a once weekly home exercise programme of 45 to 60 minutes duration. After 20 weeks, exercises are converted to home exercises, and they are monitored by a weekly sms-service. At 12 months, follow-up measurements are taken for both groups. Lymphedema is defined as 3% limb volume change from the baseline measurement.

ELIGIBILITY:
Inclusion Criteria:

* invasive unilateral breast cancer
* undergone Axillary Lymph Node Dissection (ALND), planned for Radiotherapy
* Danish speaking
* consent to participate and to be randomized to either study arm.

Exclusion Criteria:

* have undergone primary breast reconstruction
* distant metastases
* physically unable to participate for any reason
* mental illness or cognitive impairment (dementia etc.)
* no past history of lymphedema diagnosis or treatment
* not previously operated with axillary lymph node dissection either side

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2015-09; Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with Lymphedema measured by water displacement measurement | 12 months
  Lymphedema is defined as >3% increase in inter limb volume difference compared to baseline, measured by ml. water displaced by lowering arm into a tub of water.

SECONDARY OUTCOMES:
shoulder/arm/leg strength | 12 months
  change from baseline in Newtons in hand held dynometry and in 7RM tests for dynamic muscle strength.
patient reported pain | 12 months
  Pain through the study period measured on a pain scale developed to assess pain after breast cancer surgery by Gärtner et al (JAMA. 2009;302(18):1985-1992)
neuropathic pain | 12 months
  Measured by questionnaire assessment on neuropathic pain scale (NeuPPS).
Self-reported, Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-fatigue) questionnaire. | 12 months
  change from baseline in score on the FACIT-fatigue questionnaire
health related quality of life questionnaire | 12 months
  Change from baseline in Health-related quality of life Self-report, The European Organisation for Research and Treatment of Cancer (EORTC QLQ C30), breast cancer specific module (BR 23).
International Physical Activity Questionnaire (IPAQ) | baseline and 12 months
  Change in physical activity from baseline on the IPAQ
tissue composition by Dual Energy X-ray Apsorptiometry (DXA) | 12 months
  Change from baseline in tissue composition of bone mass, lean mass and fat mass, both regional and overall, assessed by Dual Energy X-ray absorptiometry (DXA).

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Oksbjerg Dalton, MD PhD, Principal Investigator — Danish Cancer Society Research Center
Locations (1):
- Danish Cancer Society Research Center, Copenhagen, Denmark